CLINICAL TRIAL: NCT04327206
Title: BCG Vaccination to Reduce the Impact of COVID-19 in Healthcare Workers (BRACE) Trial
Brief Title: BCG Vaccination to Protect Healthcare Workers Against COVID-19
Acronym: BRACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 62586; U1111-1256-4104 (Registry Identifier: The Universal Trial Number (UTN)); INV-017302 (Other Grant/Funding Number: BILL & MELINDA GATES foundation)
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Coronavirus Disease 2019 (COVID-19); Respiratory Illness; Corona Virus Infection; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BCG Vaccine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Phase III, two group, multicentre, randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The control group will receive a placebo of 0.9% sodium chloride (NaCl). Members of the research team doing the follow-up of participants and analysis will be blinded to the group allocation (by the removal of this variable and all other variables related to BCG from the dataset) until the formal detailed statistical analysis plan is confirmed and signed by all investigators and all data cleaning/preparation is complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG vaccine (Experimental): Participants will receive a single dose of BCG vaccine (BCG-Denmark). The adult dose of BCG vaccine is 0.1 mL injected intradermally over the distal insertion of the deltoid muscle onto the humerus (approximately one third down the upper arm).
  Interventions: Drug: BCG Vaccine
- 0.9% Saline (Placebo Comparator): Participants will receive a single 0.1 mL dose of 0.9%NaCl injected intradermally over the distal insertion of the deltoid muscle onto the humerus (approximately one third down the upper arm).
  Interventions: Drug: 0.9%NaCl

INTERVENTIONS:
Drug: BCG Vaccine — Freeze-dried powder: Live attenuated strain of Mycobacterium bovis (BCG), Danish strain 1331.
  Each 0.1 ml vaccine contains between 200000 to 800000 colony forming units. Adult dose is 0.1 ml given by intradermal injection
  Other Names: Bacille Calmette-Guerin Vaccine; Bacillus Calmette-Guerin Vaccine; Statens Serum Institute BCG vaccine; Mycobacterium bovis BCG (Bacille Calmette Guérin), Danish Strain 1331; BCG Denmark
  Arms: BCG vaccine
Drug: 0.9%NaCl — 0.9% Sodium Chloride Injection
  Other Names: 0.9% Saline
  Arms: 0.9% Saline

SUMMARY:
Phase III, two-group multicentre, randomised controlled trial in up to 10 078 healthcare workers to determine if BCG vaccination reduces the incidence and severity of COVID-19 during the 2020 pandemic.

DETAILED DESCRIPTION:
Healthcare workers are at the frontline of the coronavirus disease (COVID-19) pandemic. They will be randomised to receive a single dose of BCG vaccine or 0.9% NaCl placebo. Participants will be followed-up for 12 months with notification from a Smartphone application or phone calls (up to daily when ill) and surveys to identify and detail COVID-19 infection. Additional information on severe disease will be obtained from hospital medical records and/or government databases. Blood samples will be collected prior to randomisation and at 3, 6, 9 and 12 months to determine exposure to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Where required, swab/blood samples will be taken at illness episodes to assess SARS-CoV-2 infection.

The trial includes a pre-planned meta-analysis with data from 2834 participants recruited in the Stage 1 of this study, where participants were randomised to receive BCG or no BCG vaccine at the time of receiving influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Healthcare worker

  * This is defined as anyone who works in a healthcare setting or has face to face contact with patients.
* Provide a signed and dated informed consent form
* Australian sites only: If annual influenza vaccination is available, receiving the flu vaccine is an eligibility requirement. The flu vaccine will be required a minimum of 3 days in advance of randomisation in the BRACE trial.
* Pre-randomisation blood collected

Exclusion Criteria:

* Has any BCG vaccine contraindication

  * Fever or generalised skin infection (where feasible, randomisation can be delayed until cleared)
  * Weakened resistance toward infections due to a disease in/of the immune system
  * Receiving medical treatment that affects the immune response or other immunosuppressive therapy in the last year.

    * These therapies include systemic corticosteroids (≥20 mg for ≥2 weeks), non-biological immunosuppressant (also known as 'DMARDS'), biological agents (such as monoclonal antibodies against tumour necrosis factor (TNF)-alpha).
  * People with congenital cellular immunodeficiencies, including specific deficiencies of the interferon-gamma pathway
  * People with malignancies involving bone marrow or lymphoid systems
  * People with any serious underlying illness (such as malignancy)

    * NB: People with cardiovascular disease, hypertension, diabetes, and/or chronic respiratory disease are eligible if not immunocompromised, and if they meet other eligibility criteria
  * Known or suspected HIV infection,even if they are asymptomatic or have normal immune function.
  * This is because of the risk of disseminated BCG infection
  * People with active skin disease such as eczema, dermatitis or psoriasis at or near the site of vaccination
  * A different adjacent site on the upper arm can be chosen if necessary
  * Pregnant

    * Although there is no evidence that BCG vaccination is harmful during pregnancy, it is a contra-indication to BCG vaccination. Therefore, we will exclude women who think they could be pregnant or are planning to become pregnant within the next month.
    * UK specific: Although there is no evidence that BCG vaccination is harmful during pregnancy, it is a contra-indication to BCG vaccination. Therefore, we will exclude women of childbearing potential (WOCBP) who think they could be pregnant.
    * Spain specific: If the patient is female, and of childbearing potential, she must have a negative pregnancy test at the time of inclusion and practice a reliable method of birth control for 30 days after receiving the BCG vaccination.
  * Another live vaccine administered in the month prior to randomisation
  * Require another live vaccine to be administered within the month following BCG randomisation

    * If the other live vaccine can be given on the same day, this exclusion criteria does not apply
  * Known anaphylactic reaction to any of the ingredients present in the BCG vaccine
  * Previous active TB disease
  * Currently receiving long term (more than 1 month) treatment with isoniazid, rifampicin or quinolone as these antibiotics have activity against Mycobacterium bovis
* Previous adverse reaction to BCG vaccine (significant local reaction (abscess) or suppurative lymphadenitis)
* BCG vaccine given within the last year
* Have previously had a SARS-CoV-2 positive test result (positive PCR on a respiratory sample or a positive SARS-CoV-2 diagnostic antigen test approved by the local jurisdiction's public health policy)
* Already part of this trial, recruited at a different site/hospital.
* Participation in another COVID-19 prevention trial
* Have previously received a COVID-19-specific vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6828 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Symptomatic COVID-19 by 6 months | Measured over the 6 months following randomisation
  Number of participants with Symptomatic COVID-19 defined as
  * positive SARS-Cov-2 test (PCR, RAT or serology), plus
  * fever (using self-reported questionnaire), or
  * at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure (using self-reported questionnaire)
Severe COVID-19 incidence over 6 months | Measured over the 6 months following randomisation
  Number of participants with severe COVID-19 defined as:
  * positive SARS-CoV-2 test (PCR, RAT or serology), PLUS
  * death as a consequence of COVID-19, OR
  * Hospitalised as a consequence of COVID-19, OR
  * Non-hospitalised severe disease as a consequence of COVID-19, defined as non- ambulant* for ≥ 3 consecutive days unable to work** for ≥ 3 consecutive days
  (*) "pretty much confined to bed (meaning finding it very difficult to do any normal daily activities".
  (**) "I do not feel physically well enough to go to work"

SECONDARY OUTCOMES:
Symptomatic COVID-19 by 12 months | Measured over the 12 months following randomisation
  Number of participants symptomatic COVID-19 disease defined as
  * positive SARS-Cov-2 test (PCR, RAT or serology), plus
  * fever (using self-reported questionnaire), or
  * at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure (using self-reported questionnaire)
Severe COVID-19 incidence over 12 months | Measured over the 12 months following randomisation
  Number of participants with severe COVID-19 defined as:
  * positive SARS-CoV-2 test (PCR, RAT or serology), PLUS
  * death as a consequence of COVID-19, OR
  * Hospitalised as a consequence of COVID-19, OR
  * Non-hospitalised severe disease as a consequence of COVID-19, defined as non- ambulant* for ≥ 3 consecutive days unable to work** for ≥ 3 consecutive days
  (*) "pretty much confined to bed (meaning finding it very difficult to do any normal daily activities".
  (**) "I do not feel physically well enough to go to work"
Time to first symptom of COVID-19 | Measured over the 6 and 12 months following randomisation
  Participants who had either a symptomatic or severe COVID-19 episode will have time to first symptom of COVID-19 calculated as:
  [Date of any symptom onset for the first symptomatic or severe COVID-19 episode - Date of randomisation]
  Participants who have not had a symptomatic or severe COVID-19 episode will have time calculated as:
  [Earliest censoring date - date of randomisation]
Number of Episodes of COVID-19 | Measured over the 6 and 12 months following randomisation
  The total number of symptomatic or severe COVID-19 episodes (refer to outcome 3 and 4 for definitions)
Asymptomatic SARS-CoV-2 infection | Measured over the 6 and 12 months following randomisation
  Number of participants with asymptomatic SARS-CoV-2 infection defined as
  * Evidence of SARS-CoV-2 infection (by seroconversion)
  * Absence of respiratory illness (defined by trigger or non-trigger symptoms)(using self- reported questionnaire)
  * No evidence of exposure prior to randomisation
Work absenteeism due to COVID-19 | Measured within 6 and 12 months following randomisation
  Number of days (using self-reported questionnaire) unable to work (excludes quarantine/workplace restrictions) due to COVID-19 defined as
  * positive SARS-Cov-2 test (PCR, RAT or serology), plus
  * fever (using self-reported questionnaire), or
  * at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure (using self-reported questionnaire)
Bed confinement due to COVID-19 | Measured over 6 and 12 months following randomisation
  Number of days confined to bed (using self-reported questionnaire) due to COVID-19 disease defined as
  * positive SARS-Cov-2 test (PCR, RAT or serology), plus
  * fever (using self-reported questionnaire), or
  * at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure (using self-reported questionnaire)
Symptom duration of COVID-19 | Measured over 6 and12 months following randomisation
  Number of days with symptoms in any episode of illness that meets the case definition for COVID-19 disease:
  * positive SARS-Cov-2 test (PCR, RAT or serology), plus
  * fever (using self-reported questionnaire), or
  * at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure (using self-reported questionnaire)
Pneumonia due to COVID-19 | Measured over the 6 and 12 months following randomisation
  Number of pneumonia cases (using self-reported questionnaire and/or medical/hospital records) due to COVID-19
Oxygen therapy due to COVID-19 | Measured over the 6 and12 months following randomisation
  Need for oxygen therapy (using self-reported questionnaire and/or medical/hospital records) due to COVID-19
Critical care admissions due to COVID-19 | Measured over the 6 and 12 months following randomisation
  Number of admission to critical care (using self-reported questionnaire and/or medical/hospital records) due to COVID-19
Mechanical ventilation due to COVID-19 | Measured over the 12 months following randomisation
  Number of participants needing mechanical ventilation (using self-reported questionnaire and/or medical/hospital records)
Hospitalisation duration with COVID-19 | Measured over the 6 and 12 months following randomisation
  Number of days of hospitalisation due to COVID-19 (using self-reported questionnaire and/or medical/hospital records).
Mortality due to COVID-19 | Measured over the 6 and 12 months following randomisation
  Number of deaths due to COVID-19
Fever or respiratory illness | Measured over the 12 months following randomisation
  Respiratory illness using self-reported questionnaire defined as:
  * at least one sign or symptom of respiratory disease including cough, sore throat, shortness of breath, respiratory distress/failure, or runny/blocked nose (in combination with another respiratory symptom or fever).
Severe fever or respiratory illness | Measured over the 12 months following randomisation
  Severe fever or respiratory illness using self-reported questionnaire defined as:
  * Death, or
  * Hospitalised, or
  * Non-hospitalised severe disease, defined as non-ambulant1 for ≥ 3 consecutive days or unable to work2 for ≥ 3 consecutive days
Episodes of fever or respiratory illness | Measured over the 12 months following randomisation
  Respiratory illness using self-reported questionnaire defined as:
  * at least one sign or symptom of respiratory disease including cough, sore throat, shortness of breath, respiratory distress/failure, or runny/blocked nose (in combination with another respiratory symptom or fever).
Work absenteeism due to fever or respiratory illness | Measured over the 12 months following randomisation
  Number of days (using self-reported questionnaire) unable to work (excludes quarantine/workplace restrictions) due to fever or respiratory illness defined as
  * fever (using self-reported questionnaire), or
  * at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure, runny/blocked nose (using self-reported questionnaire)
Bed confinement due to fever or respiratory illness | Measured over the 12 months following randomisation
  Number of days confined to bed (using self-reported questionnaire) due to fever or respiratory illness defined as
  * fever (using self-reported questionnaire), or
  * at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure, runny/blocked nose (using self-reported questionnaire)
Symptom duration of fever or respiratory illness | Measured over the 12 months following randomisation
  Number of days with symptoms in any episode of illness that meets the case definition for fever or respiratory illness:
  * fever (using self-reported questionnaire), or
  * at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure, runny/blocked nose (using self-reported questionnaire)
Pneumonia within a febrile or respiratory illness | Measured over the 12 months following randomisation
  Number of pneumonia cases(using self-reported questionnaire and/or medical/hospital records)
Oxygen therapy for a febrile or respiratory illness | Measured over the 12 months following randomisation
  Need for oxygen therapy (using self-reported questionnaire and/or medical/hospital records)
Critical care admissions for a febrile or respiratory illness | Measured over the 12 months following randomisation
  Number of admission to critical care (using self-reported questionnaire and/or medical/hospital records)
Mechanical ventilation for a febrile or respiratory illness | Measured over the 12 months following randomisation
  Number of participants needing mechanical ventilation (using self-reported questionnaire and/or medical/hospital records)
Mortality as a consequence of an episode of fever or respiratory illness | Measured over the 12 months following randomisation
  Number of deaths
Hospitalisation duration for a febrile or respiratory illness | Measured within 6 and 12 months following randomisation
  Number of days of hospitalisation due to fever or respiratory illness (using self-reported questionnaire, medical/hospital records)
Unplanned work absenteeism for an acute illness or hospitalisation | Measured over the 6 and 12 months following randomisation
  Number of days of unplanned absenteeism for any reason (using self-reported questionnaire)
Local and systemic adverse events to BCG vaccination in healthcare workers | Measured over the 3 months following randomisation
  Adverse events (AEs), over the 3 months following randomisation, by type, severity (graded using toxicity grading scale), relationship to intervention of adverse events (AEs) of interest.
Serious Adverse Events (SAEs) to BCG vaccination in healthcare workers | Measured over the 3 months following randomisation
  SAEs over the 3 months following randomisation, by type, severity (graded using toxicity grading scale), relationship to intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Nigel Curtis, Principal Investigator — Murdoch Childrens Research Institute
Locations (36):
- Australia (13):
  - St Vincent's Hospital, Sydney, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Sydney Children's Hospital, Randwick, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Melbourne, Victoria
  - Epworth Richmond, Melbourne, Victoria
  - Monash Health- Monash Medical Centre, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Brazil (7):
  - Fundação de Medicina Tropical Dr Heitor Vieira Dourado (FMT-HVD), Manaus, Amazonas
  - Santa Casa Hospital, Campo Grande, Mato Grosso do Sul
  - CASSEMS Hospital, Campo Grande, Mato Grosso do Sul
  - Federal University of Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul
  - Hospital Regional de Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul
  - Centro de Estudos da Saúde do Trabalhador e Ecologia Humana, Rio de Janeiro, Rio de Janeiro
  - Centro de Referência Prof Hélio Fraga, Rio de Janeiro, Rio de Janeiro
- Netherlands (6):
  - Noord West Ziekenhuis, Alkmaar
  - Rijnstate Hospital, Arnhem
  - Amphia Hospital, Breda
  - St Antonius Hospital, Nieuwegein
  - Radboud UMC, Nijmegen
  - University hospital in Utrecht (UMCU), Utrecht
- Spain (5):
  - University Hospital German Trias I Pujol, Badalona, Barcelona
  - Mutua Terrassa Univeristy Hospital, Terrassa, Barcelona
  - University Hospital Cruces, Barakaldo, Bizkaia
  - Marqués de Valdecilla University Hospital, Santander
  - University Hospital Virgen Macarena, Seville
- United Kingdom (5):
  - Teign Estuary Medical Group, Teignmouth, Devon
  - Ide Lane Surgery, Alphington, Exeter
  - Travel Clinic, Exeter, Exeter
  - St Leonard's Practice, St Leonards, Exeter
  - Royal Devon and Exeter NHS Foundation Trust, Exeter

IPD SHARING:
Plan to Share IPD: Yes
Under the terms of the funding agreement with the Bill and Melinda Gates foundation, the BRACE trial has a data sharing agreement in place.
  An anonymised Individual Participant Data (IPD) dataset and a data dictionary will be provided to Vivli (https://vivli.org/) under the terms of the agreements with the Bill and Melinda Gates foundation grant and Vivli.
  After database lock, the following may be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions, under a collaborator agreement, for accessing:
  * Individual participant data that underlie the results reported in our articles after deidentification (text, tables, figures and appendices)
  * Study protocol, Statistical Analysis Plan, PICF
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After database lock, a 12-month embargo period will be in place, to allow adequate time for analyses and publication outputs. Data transfer to Vivli should occur during the embargo period.
Access Criteria: Researchers from a recognised research institution can approach MCRI for access of data.
  The researcher will need to provide evidence that the proposed use of the data has been ethically reviewed and approved by an Institutional Review Board (IRB)/ Human Research Ethics Committee(HREC), and accept MCRI's conditions, under a collaborator agreement.
URL: https://www.melbournechildrens.com/mctc/

REFERENCES:
- [Derived] Messina NL, Pittet LF, McDonald E, Moore C, Barry S, Bonten M, Byrne A, Campbell J, Croda J, Croda MG, Dalcolmo M, de Almeida E Val FF, de Oliveira RD, Dos Santos G, Douglas MW, Gardiner K, Gwee A, Jardim BA, Kollmann T, Lacerda MV, Lucas M, Lynn DJ, Manning L, Marshall H, O'Connell A, Perrett KP, Post JJ, Prat-Aymerich C, Rocha JL, Rodriguez-Bano J, Wadia U, Warris A, Davidson A, Curtis N; BRACE Trial Consortium Group. BCG vaccination of healthcare workers for protection against COVID-19: 12-month outcomes from an international randomised controlled trial. J Infect. 2024 Oct;89(4):106245. doi: 10.1016/j.jinf.2024.106245. Epub 2024 Aug 8. PMID 39127450
- [Derived] Pittet LF, Messina NL, McDonald E, Orsini F, Barry S, Bonten M, Campbell J, Croda J, Croda MG, Dalcolmo M, Gardiner K, Gwee A, Jardim B, Lacerda MVG, Lucas M, Lynn DJ, Manning L, Perrett KP, Post JJ, Prat-Aymerich C, Richmond PC, Rocha JL, Rodriguez-Bano J, Warris A, Wood NJ, Davidson A, Curtis N; BRACE Trial Consortium Group. Bacille Calmette-Guerin vaccination to prevent febrile and respiratory illness in adults (BRACE): secondary outcomes of a randomised controlled phase 3 trial. EClinicalMedicine. 2024 May 13;72:102616. doi: 10.1016/j.eclinm.2024.102616. eCollection 2024 Jun. PMID 38774675
- [Derived] Pittet LF, Moore CL, McDonald E, Barry S, Bonten M, Campbell J, Croda J, Dalcolmo M, Davidson A, Douglas MW, Gardiner K, Gwee A, Jardim B, Lacerda MVG, Lucas M, Lynn DJ, Manning L, de Oliveira RD, Perrett KP, Prat-Aymerich C, Richmond PC, Rocha JL, Rodriguez-Bano J, Warris A, Wood NJ, Messina NL, Curtis N; BRACE Trial Consortium Group. Bacillus Calmette-Guerin vaccination for protection against recurrent herpes labialis: a nested randomised controlled trial. EClinicalMedicine. 2023 Sep 11;64:102203. doi: 10.1016/j.eclinm.2023.102203. eCollection 2023 Oct. PMID 37719417
- [Derived] Pittet LF, Messina NL, Orsini F, Moore CL, Abruzzo V, Barry S, Bonnici R, Bonten M, Campbell J, Croda J, Dalcolmo M, Gardiner K, Gell G, Germano S, Gomes-Silva A, Goodall C, Gwee A, Jamieson T, Jardim B, Kollmann TR, Lacerda MVG, Lee KJ, Lucas M, Lynn DJ, Manning L, Marshall HS, McDonald E, Munns CF, Nicholson S, O'Connell A, de Oliveira RD, Perlen S, Perrett KP, Prat-Aymerich C, Richmond PC, Rodriguez-Bano J, Dos Santos G, da Silva PV, Teo JW, Villanueva P, Warris A, Wood NJ, Davidson A, Curtis N; BRACE Trial Consortium Group. Randomized Trial of BCG Vaccine to Protect against Covid-19 in Health Care Workers. N Engl J Med. 2023 Apr 27;388(17):1582-1596. doi: 10.1056/NEJMoa2212616. PMID 37099341
- [Derived] Pittet LF, Messina NL, Gardiner K, Orsini F, Abruzzo V, Bannister S, Bonten M, Campbell JL, Croda J, Dalcolmo M, Elia S, Germano S, Goodall C, Gwee A, Jamieson T, Jardim B, Kollmann TR, Guimaraes Lacerda MV, Lee KJ, Legge D, Lucas M, Lynn DJ, McDonald E, Manning L, Munns CF, Perrett KP, Prat Aymerich C, Richmond P, Shann F, Sudbury E, Villanueva P, Wood NJ, Lieschke K, Subbarao K, Davidson A, Curtis N; BRACE trial Consortium Group. BCG vaccination to reduce the impact of COVID-19 in healthcare workers: Protocol for a randomised controlled trial (BRACE trial). BMJ Open. 2021 Oct 28;11(10):e052101. doi: 10.1136/bmjopen-2021-052101. PMID 34711598
- [Derived] Crisan-Dabija R, Grigorescu C, Pavel CA, Artene B, Popa IV, Cernomaz A, Burlacu A. Tuberculosis and COVID-19: Lessons from the Past Viral Outbreaks and Possible Future Outcomes. Can Respir J. 2020 Sep 5;2020:1401053. doi: 10.1155/2020/1401053. eCollection 2020. PMID 32934758